CLINICAL TRIAL: NCT06006676
Title: Mechanical Ventilation to Accelerate Recovery of Lung Function in Veno-venous Extracorporeal Membrane Oxygenation; Lung Rest Or Moderate Mechanical Ventilation in ECMO: Randomized Trial
Brief Title: IMV to Accelerate Recovery of Lung Function in Veno-venous Extracorporeal Membrane Oxygenation; Lung Rest Or Moderate Mechanical Ventilation in ECMO
Acronym: ROMEO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 256932
Record Dates: First submitted 2021-10-06; First posted 2023-08-23 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: ARDS
Keywords: ARDS; Critical Care; ECMO

STUDY DESIGN:
Intervention Model Description: Parallel group randomised prospective open label trial of two ventilation strategies during V-V ECMO for ARDS with standardised crossover weaning studies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Near Apnoeic Ventilation (Experimental): Near Apnoeic ventilation (with a respiratory rate of 2 breaths per minute, plateau pressure of 30cmH20 and PEEP set according to the mean airway pressure being delivered during mechanical ventilation prior to randomisation) for a 72 hour period following randomisation
  Interventions: Other: Near Apnoeic ventilation; Other: Crossover standardised ECMO weaning trials
- Standard Care (Active Comparator): Standard care for patient on ECMO as per consultant with respiratory rate of 15-30, PEEP of 10cmH20 or more and Plateau pressure of 25cmH20 or less for a 72 hour period following randomisation
  Interventions: Other: Crossover standardised ECMO weaning trials

INTERVENTIONS:
Other: Near Apnoeic ventilation — Near Apnoeic ventilation (with a respiratory rate of 2 breaths per minute, plateau pressure of 30cmH20 and PEEP set according to the mean airway pressure being delivered during mechanical ventilation prior to randomisation) for a 72 hour period following randomisation
  Arms: Near Apnoeic Ventilation
Other: Crossover standardised ECMO weaning trials — When all patients are eligible for a trial of ECMO weaning, they will have standardised ECMO weaning trials lasting up to 1 hour with 0 sweep gas flow. 1) "One-stage weaning"- sweep gas flow rate sequentially decreased to zero 2) "Two-stage weaning"- fraction of oxygen of sweep gas flow decreased to 0.21 sequentially. Then the sweep gas flow rate decreased to 0 sequentially

SUMMARY:
Feasibility trial to inform a future multicentre randomized control trial. The investigators aim to evaluate the feasibility of a trial of near apnoeic ventilation (two breaths per minute) compared with standard ventilation (respiratory rate between 10 and 30 breaths) for patients with acute respiratory distress syndrome (ARDS) supported with veno-venous extracorporeal membrane oxygenation (V-V ECMO). Additionally, when a patient is determined as ready to wean from ECMO the investigators will explore the feasibility of two ECMO weaning strategies and explore the physiological effects on respiratory effort and gas exchange.

DETAILED DESCRIPTION:
Background

Acute respiratory distress syndrome (ARDS) is a common clinical syndrome characterised by life threatening respiratory failure requiring mechanical ventilation. Although lifesaving, mechanical ventilation can cause further injury to the lungs, known as ventilator-induced lung injury (VILI). Strategies to mitigate VILI in ARDS have proven to improve patient outcomes. ARDS patients that have severe lung failure, despite mechanical ventilation, often require veno-venous extracorporeal membrane oxygenation (ECMO). ECMO uses an artificial membrane lung to take over gas exchange. This allows reduction in injurious ventilator settings thereby also reducing VILI.

While the indications for ECMO initiation are standardised in the UK and ECMO utilisation is increasing,there remains uncertainty as to the best approach to mechanical ventilation whilst patients are receiving ECMO and what strategies are maximally attenuating VILI during its use. Importantly it is known that despite the reduction in ventilatory pressures and volumes facilitated by ECMO, these sickest and most fragile lungs continue to be susceptible to VILI. A reduction in respiratory rate (RR) to near apnoeic ventilation (2 breaths per minute) seems to be associated with the greatest physiological reduction in VILI components, whilst maintaining important physiological mechanisms such as surfactant production which rely on some lung inflation. Employing a near apnoeic ventilation strategy may be associated with faster resolution of ARDS resulting in reduced duration of ECMO, ventilation and ICU stay, and healthcare costs.

Rationale

Interventions which mitigate VILI lead to less lung inflammation/oedema and better outcomes in ARDS patients. However, the recent REST trial of extracorporeal carbon dioxide removal showed that the resultant modest reduction in volume and pressure had no clinical effect. Hence, a modest reduction in ventilation may not be as effective as an almost complete absence (near apnoeic) of ventilation. The latter can only be achieved alongside ECMO support. Reductions in respiratory rate to near apnoeic ventilation have multiple effects on VILI, including:

1. Modulation of disease activity through reduced opening and closing of lung units (atelectrauma);
2. Reductions in frequency of applied driving pressure and overall intensity of minute ventilation (barotrauma)
3. Prevention of overdistension of the aerated lung (volutrauma)
4. Attenuation of circulating markers of lung injury and inflammation ('biotrauma')
5. Reduced development of aberrant fibrosis within the lung [9]. Patients on ECMO are prone to pulmonary fibrosis, for which VILI is known to be major contributor

Multinational surveys of mechanical ventilation during ECMO support show that 45.7% of centres used a moderate respiratory rate (10-20 breaths per minute) delivered with ~10-15 cmH2O PEEP and 10-15 cmH2O driving pressure. Evidence shows a 3% increase in the hazard of death for every 1 cmH2O increase in ventilator driving pressure during ECMO support. Taken together, international experience and trend show that ventilator mechanical power (a measure of the energy transmitted to the lung) is a major determinant of VILI and is only modestly decreased by the currently employed moderate ventilation strategies which mainly reduce the driving pressure applied per breath. Mechanical power is, however, significantly reduced by lower respiratory rates. Near apnoeic ventilation during ECMO is clinically feasible with gas exchange and oxygen delivery being maintained by ECMO.

The ROMEO trial

The investigators have conducted a detailed search of PubMed, Ovid, Cochrane databases, Google Scholar and the WHO International Clinical Trials Registry Platform. To-date, no large prospective studies have or are addressing the use of near apnoeic ventilation during ECMO. Consequently, a multicentre randomised open label study of near apnoea ventilation versus standard of care is planned. This future multicentre trial will be powered for patient centred outcomes (e.g., time to ECMO decannulation and mortality) together with a trial cost utility analysis at 12 months.

To demonstrate the feasibility of our trial design, we will conduct a 50 patient feasibility study at Guy's and St Thomas' NHS Foundation Trust. This will evaluate the feasibility of the intervention (ability to recruit; ability to deliver the ventilator strategy; ability to deliver the ECMO weaning strategies), the physiological changes induced by near apnoea ventilation together with the impact on plasma and broncho-alveolar lavage biomarkers and collect exploratory data on clinical outcomes.

As there is a paucity of evidence regarding predictors of ECMO weaning success, we will evaluate comprehensive physiological data obtained during each weaning trial attempt to evaluate the patient-ventilator-membrane lung interactions.

ELIGIBILITY:
Inclusion criteria

* Adult patients aged 18 years or older on the date of screening
* Acute and potentially reversible cause of ARDS
* Receiving invasive mechanical ventilation
* Requiring ECMO for severe ARDS
* Tidal volume ≥ 2.5ml/kg predicted body weight

Exclusion criteria:

Patients who meet the one or more of the following will be excluded from the trial.

* Declined consent
* >12 hours following ECMO initiation
* Patient likely to die or for withdrawal of life sustaining therapies within 24 hours
* Use of V-A ECMO or hybrid ECMO modes
* Current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients receiving a ventilation strategy other than the assigned ventilation strategy over the 72 hour period following randomisation | During the 72 hours following randomisation
  Number of patients receiving a ventilation strategy other than the assigned ventilation strategy over the 72 hour period following randomisation (excluding time off the ICU for imaging or surgical/interventional procedures)

SECONDARY OUTCOMES:
Time to achieving carbon dioxide output (VCO2) natural lung > 50% of total of CO2 output | Up to 6 months following date of randomisation
  Time to achieving carbon dioxide output (VCO2) natural lung > 50% of total of VCO2 (VCO2 from ECMO plus VCO2 from natural lung)
Time to achieve a PaO2 > 30 kPa with Cilley's test (arterial oxygenation achieved after an increase in FiO2 to 1.0 with no other changes to the ventilator or ECMO settings) | Up to 6 months following date of randomisation
  Time to achieve a PaO2 > 30 kPa with Cilley's test (arterial oxygenation achieved after an increase in FiO2 to 1.0 with no other changes to the ventilator or ECMO settings)
Rate of successful ECMO weaning trial | Up to 6 months following date of randomisation
  Proportion of ECMO weaning trials which result in success (sweep gas flow of 0 for 1 hour without: respiratory rate >35, P0.1 measured by ventilator less than -10cmH2O, oxygen saturations <88%, pH <7.35 due to increasing PaCO2, obvious clinical distress)
Number of patients with non-adherence to assigned ECMO weaning strategy | Up to 6 months following date of randomisation
  Number of patients in whom there is non-adherence to the assigned ECMO weaning strategy (for example, clinicians make a decision to decannulate despite the outcome of a weaning trial)
Change in total compliance of the respiratory system during a low flow pressure volume loop after 72hrs of the assigned ventilation strategy | 72 hours
  Difference between 72 hour and baseline total compliance of the respiratory system (compliance of the whole pressure volume loop curve obtained with 8L/s flow, pressure from 5 to 40cmH2O with volume limit of 12mls/kg ideal body weight

OTHER OUTCOMES:
Time from randomisation to ECMO decannulation | Up to 6 months following date of randomisation
  Time from randomisation to ECMO decannulation
Rate of decannulation from ECMO | Up to 6 months following date of randomisation
  Rate of decannulation from ECMO
Time to achieve a successful ECMO weaning trial | Up to 6 months following date of randomisation
  Time to achieve a successful ECMO weaning trial
Duration of invasive mechanical ventilation and total ventilator days (excluding high-flow nasal cannulae) | Up to 6 months following date of randomisation
  Duration of invasive mechanical ventilation and total ventilator days (excluding high-flow nasal cannulae)
Length of stay in the ECMO centre | Up to 6 months following date of randomisation
  Length of stay in the ECMO centre
ECMO mortality | Up to 6 months following date of randomisation
  Mortality at the ECMO centre
Change in oxygen saturations during a weaning trial | Up to 6 months following date of randomisation
  Difference between baseline and end of trial value of oxygen saturations derived from pulse oximetry
Change in oesophageal pressure swing during a weaning trial | Up to 6 months following randomisation
  Difference between baseline and end of trial value of oesophageal pressure swing
Change in ventilatory efficiency during a weaning trial | Up to 6 months following randomisation
  Difference between baseline and end of trial value of ventilatory efficiency, calculated as the minute ventilation (measured by mechanical ventilator) divided by the CO2 clearance by the natural lung (measured using volumetric capnography)
Change in modified Borg Dyspnoea Score during a weaning trial | Up to 6 months following randomisation
  Difference between baseline and end of trial modified Borg dyspnoea score
Change in haematocrit during a weaning trial | Up to 6 months following randomisation
  Difference between baseline and end of trial haematocrit measured on an arterial blood gase

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Camporota, MD, PhD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guys & St. Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No